CLINICAL TRIAL: NCT00059826
Title: A Phase II Study of Interferon-Based Adjuvant Chemoradiation in Patients With Resected Pancreatic Adenocarcinoma
Brief Title: Adjuvant Chemoradiotherapy and Interferon Alfa in Treating Patients With Resected Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z05031; CDR0000298776 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Introns; Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interferon-based chemoradiation therapy (Experimental): Cycle 1: Chemoradiotherapy (CRT)
  * 5-fluorouracil continuous infusion (CI) via an ambulatory infusion pump into a central venous catheter at 175 mg/m2/day for 38 consecutive days, unless toxicity occurs
  * cisplatin given on the first day only of each week of this cycle (days 1, 8, 15, 22, 29, 36)
  * IFN-alpha-2b 3 million units given subcutaneously on days 1, 3, and 5 of each week for 5½ weeks
  * XRT 5040 cGy total, in 28 fractions, at 180 cGy/fraction daily, Monday - Friday, for 5½ weeks
  Cycles 2 and 3: Post-CRT Chemotherapy
  Post-CRT chemotherapy starts 4 - 6 weeks after completion of Cycle 1, unless the study physician deems further delay is necessary. Patients will be given 2 cycles of chemotherapy (cycles 2 and 3).
  -- 5-fluorouracil continuous infusion via an ambulatory infusion pump into a central venous catheter at 200 mg/m2/day for 6 weeks followed by 2 weeks of rest
  Interventions: Biological: interferon-alfa-2b; Drug: cisplatin; Drug: 5-fluorouracil; Radiation: radiation therapy

INTERVENTIONS:
Biological: interferon-alfa-2b — IV
  Other Names: IFN-alpha-2b
Drug: cisplatin — IV
Drug: 5-fluorouracil — IV
  Other Names: 5-FU
Radiation: radiation therapy
  Other Names: XRT

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of tumor cells. Radiation therapy uses high-energy radiation from x-rays and other sources to kill tumor cells. Combining chemotherapy with interferon alfa and giving them with radiation therapy after surgery may kill any remaining tumor cells.

PURPOSE: Phase II trial to study the effectiveness of adjuvant chemoradiotherapy and interferon alfa in treating patients who have resected stage I, stage II, or stage III pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the disease-free and overall survival of patients with resected pancreatic adenocarcinoma treated with adjuvant chemoradiotherapy comprising fluorouracil, cisplatin, and interferon alfa.
* Determine the rate and severity of acute and late toxic effects in patients treated with this regimen.
* Determine the local-regional disease control and distant disease control in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Chemoradiotherapy (CRT): Patients receive fluorouracil IV continuously on days 1-38; cisplatin IV over 1 hour on days 1, 8, 15, 22, 29, and 36; and interferon alfa subcutaneously on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, 33, 36, and 38. Patients also undergo radiotherapy on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-38.
* Post-CRT chemotherapy: Beginning 4-6 weeks after the completion of CRT, patients receive fluorouracil IV continuously on days 1-42. Treatment repeats every 56 days for a total of two courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 2 years, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be > 18 years of age.
2. Patient must have a documented ECOG/Zubrod performance status of 0 or 1, within 7 days prior to registration.
3. Patient must have pathological stage T1-3, N0-1, M0 adenocarcinoma of the head of the pancreas according to the American Joint Committee on Cancer (AJCC) staging system.

   * NOTE: The pathology report must be submitted to ACOSOG on the Pathology Report Shuttle CRF.
4. Patient must have undergone a potentially curative gross total resection by pancreaticoduodenectomy (includes R0 [no residual tumor] or R1 [microscopic residual tumor]) within 56 days prior to beginning treatment. NOTE: The operative report must be submitted to ACOSOG on the Operative Report Shuttle CRF.
5. Patient must have stable or increasing weight in the 14 days prior to the start of treatment, otherwise supplemental nutrition (e.g. feeding jejunostomy, PEG, TPN) must be initiated prior to the start of treatment.6. Patient must have adequate bone marrow, hepatic and renal function, within 7 days prior to registration:

   * WBC > 3,000 mm^3
   * ANC > 1,500 mm^3
   * hemoglobin > 9.5 mg/dl
   * platelet count > 100,000 mm^3
   * total bilirubin < 3 mg/dl
   * AST (SGOT) < 2.0 times institutional upper limit of normal (ULN)
   * ALT (SGPT) < 2.0 times institutional ULN
   * alkaline phosphatase < 2.0 times institutional ULN
   * serum creatinine < 1.5 times institutional ULN

7. Patient must have a baseline diagnostic CT scan of the chest and CT scan with IV contrast (or MRI) of abdomen/pelvis, within 30 days prior to registration, to exclude metastatic disease.

8. If female of childbearing potential, patient must have a negative urine or serum pregnancy test, within 7 days prior to registration. NOTE: Postmenopausal women must have been amenorrheic for at least 12 consecutive months to be considered not of childbearing potential.

9. Patient (male or female) of reproductive potential must agree to use medically acceptable contraception during the study. NOTE: Medically acceptable contraceptives include: (1) surgical sterilization, (2) approved hormonal contraceptives (such as birth control pills, Depo-Provera, or Lupron Depot), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD).

10. Patient, or the patient's legally acceptable representative, must sign and date an informed consent PRIOR to registration and the performance of any study related procedures.

11. Patient, or the patient's legally acceptable representative, must provide written authorization to allow the use and disclosure of their protected health information.

- NOTE: This may be obtained in either the study-specific informed consent or in a separate authorization form and must be obtained from the patient prior to study registration.

12. If patient is a cancer survivor, all of the following criteria must be met and documented in the patient's medical record:

1. Patient has undergone potentially curative therapy for all prior malignancies.
2. No evidence of prior malignancies for at least 5 years (except for successfully treated cervical carcinoma in situ, lobular carcinoma in situ of the breast, or nonmelanoma skin cancer).
3. No evidence of recurrence of any prior malignancy.

Exclusion Criteria:

1. Patient has pancreaticoduodenectomy histopathology of adenosquamous carcinoma, ampullary carcinoma, carcinoid tumor, cystadenocarcinoma, cystadenoma, distal common bile duct carcinoma, duodenal carcinoma, or islet cell carcinoma.
2. Patient is pregnant or lactating.
3. Patient has recurrent pancreatic cancer.
4. Patient has received prior systemic chemotherapy or radiotherapy for pancreatic cancer.
5. Patient has received external beam photon (x-ray) therapy to the chest, abdomen or pelvis.
6. Patient has received any biologic/ immunologic therapies.
7. Patient has received chronic immunotherapy (e.g. prednisone or methotrexate) for collagen vascular disease or other chronic immunologic abnormality.
8. Patient has a preexisting psychiatric condition, especially depression, or a history of severe psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2003-03; Primary Completion 2007-07 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Overall survival at 18 months | at 18 months

SECONDARY OUTCOMES:
Toxicity | at 18 months
Disease-free survival | at 18 months
Local-regional disease control | at 18 months
Distant disease control | at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincent J. Picozzi, MD, Study Chair — Floyd & Delores Jones Cancer Institute at Virginia Mason Medical Center
Locations (14):
- United States (14):
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Picozzi VJ, Abrams RA, Decker PA, Traverso W, O'Reilly EM, Greeno E, Martin RC, Wilfong LS, Rothenberg ML, Posner MC, Pisters PW; American College of Surgeons Oncology Group. Multicenter phase II trial of adjuvant therapy for resected pancreatic cancer using cisplatin, 5-fluorouracil, and interferon-alfa-2b-based chemoradiation: ACOSOG Trial Z05031. Ann Oncol. 2011 Feb;22(2):348-54. doi: 10.1093/annonc/mdq384. Epub 2010 Jul 29. PMID 20670978
- [Result] Picozzi VJ, Abrams RA, Traverso LW, et al.: ACOSOG Z05031: initial report of a multicenter, phase II trial of a novel chemoradiation protocol using cisplatin, 5-FU, and alpha- interferon as adjuvant therapy for resected pancreas cancer. [Abstract] American Society of Clinical Oncology 2008 Gastrointestinal Cancers Symposium, 25-27 January 2008, Orlando, FL. A-125, 2008.
- [Result] Picozzi VJ, Abrams RA, Traverso LW, et al.: ACOSOG Z05031: report on a multicenter, phase II trial for adjuvant therapy of resected pancreatic cancer using cisplatin, 5- FU, and alpha-interferon. [Abstract] J Clin Oncol 26 (Suppl 15): A-4505, 2008.